



### MAIN INFORMED CONSENT FORM

Title of the Study: Adaptive evaluation of mHealth and conventional adherence

support interventions to optimize outcomes with new treatment regimens for drug-resistant tuberculosis and HIV in South

Africa (ADAP-TIV)

**Sponsor:** Centre for AIDS Programme of Research in South Africa

(CAPRISA)

**Funder:** U.S. National Institute of Health

Principal Investigators: Dr. Kogieleum Naidoo

Dr. Max O'Donnell

## Dear Patient

You are being invited to take part in this research study because you are eligible for a **study on engagement in care for drug resistant tuberculosis and HIV**. The doctor in charge of this study is Dr. Kogieleum Naidoo. You are being asked to take part in this study because you are HIV positive and on ART and have been recently diagnosed with drug-resistant tuberculosis and will be starting treatment. Before you decide if you want to enroll in this study, we want you to know about the study.

This consent form gives you information about this study, which will be done at King DinuZulu Hospital Complex. Please ask questions and discuss any concerns you may have with the research staff. If you agree to take part in this study, you will be asked to sign this consent form. You will be given a copy of this consent form to keep.

### Please note that:

- Your participation in this study is entirely voluntary. You may decide not to participate in the study, but you will still receive the same medical care as determined by your doctor.
- You may stop taking part in the study at any time and this will not affect the care you receive at the hospital.
- You may contact the Biomedical Research Ethics Committee (BREC) on 031-260 4769 or 031-260 1074 (business hours) if you have questions about your rights as a research subject.

### WHY IS THIS STUDY BEING DONE?

The purpose of this study is to help doctors understand the benefit of a new program to improve adherence to TB and HIV medicines. 'Adherence' to your medicines refers to how well you take your TB and HIV medicines as prescribed by the doctor. Taking all your medication will help kill





the bugs causing your TB. Taking medication for TB is the most important thing that will determine if you get better and live longer. By allowing us to ask questions, collect information, and collect periodic sputum and blood samples from you we will be able to assess the effectiveness of programs to increase medication adherence and its relationship with treatment outcomes for drug-resistant tuberculosis.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Approximately 360 participants will take part in this study.

#### WHAT IS INVOLVED IN THIS STUDY?

You will be assigned to one of four treatment groups by random choice. Randomization is like a coin flip. We do not control to which group you will be assigned. The entire study will last until you complete your tuberculosis treatment or one year, whichever is longer.

In each group, you will continue to come to the clinic for monthly visits until 6 months have passed since you enrolled into the study. You will also return to the clinic for a follow-up visit at 12 months following enrollment. We will schedule a telephonic visit when you complete your TB treatment, which typically happens between 6-18 months following treatment start.

Each group will receive an enhanced standard of care, but there are four different versions of the program in which you will participate. You will not know which version of the program you are receiving.

If you would like to participate in this study, you will be asked questions about your medical history and any medicines that you have taken. If you agree to participate in the study, we will collect medical information including blood test results, X-rays and sputum results. These tests will include HIV test results, test to check how many cells you have in your body to fight infections (CD 4 T cell counts), and tests to check how many copies of HIV you have in your blood (viral load tests), if applicable. In addition to your regularly scheduled clinical visits, we will ask you to produce two sputum samples and provide a blood sample (at the Enrollment visit, months 2, 6, and 12).

As part of the study, you may be asked to participate in one-on-one counseling sessions at each clinic visit. You may also be asked to participate in counseling sessions before being discharge from the hospital.

### Adherence

We may ask questions to assess how well you take your medication. Depending on the group into which you are randomized you may be given an electronic pillbox which will count the number of pills taken.





# Adherence Support Groups

In addition to the clinic visits, you may be asked to participate in a patient support discussion group that is about an hour long, which will happen at least once a month. This discussion group is to help you identify challenges for your treatment and get support from other patients who are taking similar treatment. These sessions will be audio-recorded.

## Use of Data/Specimens

For this study we may share your sputum and blood samples with other researchers at other institutions (including collaborators at Columbia University in New York, USA) so that other research studies can be done now or in the future. If your samples are shared with other institutions, your identifying information will not be included. If you agree to let us keep your samples for future research, your samples will be stored at the CAPRISA Research Laboratory for 10 years. If we are required to perform any additional tests on your samples, CAPRISA will contact the Biomedical Research Ethics Committee for approval. There will be no additional medications given to you, other than the standard medications your doctors prescribe for you.

Some research using tissue allows the researchers to make medical tests or treatments that may have commercial value. If this happens, there are no plans to pay you for any products or treatments that are made, or for using your samples.

## Telephonic Contact and Optional Home Visits

Study staff may contact you on your cell phone or home phone to discuss your treatment and/or progress. Study staff may also contact you about the study by text message. Study staff will ask you to go to a quiet place where you cannot be disturbed so you may answer confidential questions.

The study staff may decide to visit you at your home to discuss the study and the care you are receiving for your drug-resistant TB and HIV. If you are given an electronic pill box, study staff may want to visit your home to discuss the pillbox and to be sure it is working properly. If a member of the study staff would like to visit you at home, you will be contacted at home to determine a date and time that works for you. We will take measures to ensure that the reason for

| our visit remains confidential. | | |
|---|---|---|
| By agreeing to participate in this studecide not to participate in potential | | , , |
| HOME VISITS (Initial your resp | onse) | |
| YES, I agree to home vis | sits | |
| NO, I do not agree to hor | me visits | |
| ADAP-TIV<br>Version 1.0 | Page 3 of 8 | 08 April 2022 |





### HOW LONG WILL I BE IN THE STUDY?

You will be followed through the course of your drug-resistant tuberculosis treatment (normally between 6-18 months).

## WHAT ARE THE POTENTIAL RISKS ASSOCIATED WITH THIS STUDY?

# Loss of confidentiality

A risk of taking part in this study is the possibility of a loss of confidentiality. Loss of confidentiality includes having your personal information shared with someone who is not on the study team and was not supposed to see or know about your information. The study team plans to protect your confidentiality.

## Psychological risk

There is a potential risk for psychological distress from the questions that will be asked regarding the barriers to adherence. Should you feel uncomfortable at any point, please inform one of the study staff. Please also take care not to disclose information you are not comfortable sharing, and please note that you can withdraw from the study at any time.

### WHAT ABOUT CONFIDENTIALITY?

Your medical records, personal information, and the results of your HIV tests and other medical and laboratory evaluations will be kept strictly confidential within the extent of South African law. Only your doctor and/or study staff will know the results of your tests. The study research team will give you a unique number once you are enrolled into the study. A different number will be given for each participant in the study. This unique number and not your name (or any other information that could be used to identify you) will be used for all of your study-related records. Any publication of this study will not use your name or identify you personally.

Every effort will be made to protect your confidentiality but we cannot guarantee absolute confidentiality. The study team plans to protect your confidentiality. However, your confidentiality cannot be assured in adherence support groups discussions. While we will inform participants to respect each other's confidentiality, we cannot guarantee that participants will do so. You should thus be careful what you disclose in these adherence support group sessions.

Your specimens, information from medical records, and questionnaire responses will be assigned a code number, and separated from your name or any other information that could identify you. The research file that links your name to the code number will be kept in a locked file cabinet or an encrypted data file and only the investigator, study staff and monitors/sponsor representatives will have access to the file.

Your personal information may be disclosed if required by law. Your records may also be reviewed by regulatory authorities, the Ethics Committees and study staff.





### ARE THERE BENEFITS TO TAKING PART IN THIS STUDY?

If you participate in this study, there may or may not be a direct benefit to you. The goal of this study is to improve outcomes by delivering enhanced care. There is no guarantee of a direct benefit received by taking part in this study. However, the knowledge gained may guide investigators in improving treatment support and programs for individual patients in the current study and in the future.

It is important to note that there are no significant risks or benefits for you to produce a sputum sample.

## WHAT OTHER CHOICES DO I HAVE BESIDES THIS STUDY?

If you choose not to participate in this study, you can still receive medical treatment at King DinuZulu referral hospital or your referring local clinic.

## REIMBURSEMENT

You will be compensated R150 for each study visit for your time and effort provided in participating in the research. For the follow-up visits you will also be compensated R150. For study team initiated interim visits you will be compensated R150.

### WHAT ARE THE COSTS TO ME?

Taking part in this study will not involve additional costs to you. Treatment for drug resistant TB and HIV is provided at no cost according to the practices and policies of King DinuZulu referral hospital and the KwaZulu-Natal Department of Health.

## **ALTERNATIVES**

Taking part in this study is your choice. You may choose to either take part or not take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care.

If you have any questions while taking part in this research study, you should contact the Principal Investigator:

Dr. Kogieleum Naidoo

Telephone: +27 31 655 5707 Email: kogie.naidoo@caprisa.org





For questions about your rights as a research participant, or any problems related to the study you may contact:

## **Biomedical Research Ethics Committee (BREC)**

Research Office, Westville Campus Govan Mbeki Building Private Bag X 54001 Durban 4000 KwaZulu-Natal, SOUTH AFRICA

Tel: +27 31 260 4769 (business hours) - Fax: +27 31 2604 609

Email: BREC@ukzn.ac.za

Your participation in this research is voluntary, and you will not be penalized or lose benefits if you refuse to participate or decide to stop.

If you agree to participate, you will be given a signed copy of this document.

The research study, including the above information, has been described to me orally. I understand what my involvement in the study means and I voluntarily agree to participate.

It is possible that in the future a genetic test could be done on your stored samples.

| Name of Participant | Signature of Participant | Date dd/mmm/yy |
|---|---|---|
| Name of Witness<br>(Where applicable) | Signature of Witness | Date dd/mmm/yy |
| Name of Study Staff | Signature of Study Staff | Date dd/mmm/yy |





### **USE OF STORED SAMPLES**

Samples will be collected and stored for future research use. For this study we may share your sputum and blood samples with other researchers at other institutions (including collaborators at Columbia University in New York, USA) so that other research studies can be done now or in the future. If your sputum samples are shared with other institutions, your identifying information will not be included. The research team may use these samples to confirm test results or to do additional new tests if required. Your samples will not be sold or used in other products that make money for researchers. Should you decide not to have your samples stored this will not affect your ability to take part in the study. Your decision will not affect the quality of care you receive at the clinic.

To protect your identity your sample container will not have your name or any information that may identify you. Only your study number will be used on sample containers. If you do not agree, then samples for storage will not be collected. If you agree now and later change your mind, your sample will not be used for future testing. No matter what you decide, it will not affect your participation in the study and this will not affect the quality of care you receive from study staff.

| <br>YES, I agree to have my samples stored |
|---------------------------------------------------|
| <br>NO, I do not agree to my samples being stored |

Any studies that use your samples will be reviewed by the Biomedical Research Ethics Committee of the University of KwaZulu-Natal.

The researchers do not plan to contact you or your regular doctor with any results that are done on the stored samples after the study has been completed.

This is because research tests are often done with experimental procedures so the results from one study are generally not useful for making decisions on managing your health. Should a rare situation come up where the researchers decide that a specific test result would provide important information for your health, the researchers will notify the study doctor who will try to contact you or your regular doctor. If you wish to be notified of this type of test result, you need to make sure that you contact the study nurse or doctor with any changes to your phone number or address. If you want your regular doctor to be told about this kind of test result, you need to provide the study team with the contact details of your regular doctor.





| Name of Participant | Signature of Participant | Date dd/mmm/yy |
|---|---|---|
| I give my permission for<br>South Africa. | any collected samples to be shipp | oed to collaborators outside of |